CLINICAL TRIAL: NCT05022615
Title: Comparison of Standard and Ultrawide Field Imaging Systems
Brief Title: Comparing 3 Imaging Systems
Acronym: COCO
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0977; A536000 (Other: University of Wisconsin-Madison); Protocol Version 4-22-2021 (Other: University of Wisconsin-Madison)
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (4):
- Mild Non-Proliferative Diabetic Retinopathy (NPDR): Presence of at least one retinal microaneurysm or hemorrhage as determined by clinician.
  Interventions: Diagnostic Test: Topcon Camera; Diagnostic Test: Optos Camera; Diagnostic Test: Clarus Camera
- Moderate NPDR: Increasing hemorrhages and microaneurysms as well as cotton wool spots, venous beading (VB) or Intraretinal microvascular abnormalities (IRMA) to a mild degree as determined by clinician
  Interventions: Diagnostic Test: Topcon Camera; Diagnostic Test: Optos Camera; Diagnostic Test: Clarus Camera
- Severe NPDR: "4-2-1" rule-that is, one has severe NPDR if hemorrhages or microaneurysms, or both, appear in all four retinal quadrants; venous beading appears in two or more retinal quadrants; or prominent IRMAs are present in at least one retinal quadrant as determined by clinician.
  Interventions: Diagnostic Test: Topcon Camera; Diagnostic Test: Optos Camera; Diagnostic Test: Clarus Camera
- Proliferative Diabetic Retinopathy (PDR): Neovascularization, either on or within one disc diameter (DD) of the optic disc (NVD) or elsewhere in the retina (NVE); a preretinal hemorrhage (PRH); or vitreous hemorrhage (VH) as determined by the clinician.
  Interventions: Diagnostic Test: Topcon Camera; Diagnostic Test: Optos Camera; Diagnostic Test: Clarus Camera

INTERVENTIONS:
Diagnostic Test: Topcon Camera — Standard 7 field imaging
Diagnostic Test: Optos Camera — Ultrawide field imaging
Diagnostic Test: Clarus Camera — Ultrawide field imaging

SUMMARY:
The purpose of this study is to evaluate the quality of ocular images captured on 3 different cameras of patients with diabetic retinopathy. The study will determine whether diabetic retinopathy assessment is comparable between the cameras. The research is being done to see if a camera takes higher quality pictures over the other cameras.

60 participants will be enrolled into this study. Participants need to have diabetic eye disease. This is a one-time study visit that lasts approximately 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* any race
* Established diagnosis of diabetes.
* Willing to participate as evidenced by signing the written informed consent.

Exclusion Criteria:

* Unable to tolerate ophthalmic imaging.
* Ocular is media not sufficiently clear to obtain technically acceptable ultrawide field images.
* History of panretinal laser photocoagulation or vitrectomy (history of anti-vascular endothelial growth factor treatment is not an exclusion criteria).
* Presences of confounding abnormalities such as age-related macular degeneration, retinal vein occlusion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (18 or older) with either Type 1 or Type 2 diabetes presenting at a single center of an ophthalmic retina practice for examination of diabetic retinopathy including color photography for standard medical care.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Early Treatment Diabetic Retinopathy Study (ETDRS) Severity Level within the 7 standard fields of Clarus, Optos, and Standard 7 Field imaging and statistical comparison | 1 day
  The images captured within the 7 standard fields on each camera will be graded using the ETDRS severity scale. The total range of possible scores for severity level is from 10 (no DR) to 80 (PDR with vitreous hemorrhage); higher scores indicate increasing severity.
  Details of ETDRS severity scale: 10-No DR, 15-Probable DR, no MAs, 20-MAs only, 35-Mild NPDR, 43,47-Moderate NPDR, 53-Severe NPDR, 60-PDR status post scatter photocoagulation, 61,65,71-PDR, 80-PDR with vitreous hemorrhage, 90,95-Ungradable.
  ETDRS level agreement will be cross-tabulated and κ statistics calculated and assessed: <0.20, poor; 0.21-0.40, fair; 0.41-0.60, moderate; 0.61-0.80, substantial; and 0.81-1.00, almost perfect strength of agreement. Unweighted κ will be used to avoid potential bias by weighting. Agreement will also be tested for each severity level and k statistics analyzed.
Number of Ungradable ETDRS Images within the 7 standard fields of Clarus, Optos, and Standard 7 Field imaging | 1 day
  The images captured within the 7 standard fields on each camera will be graded using the ETDRS severity scale. The proportion of ungradable images will be documented. On all tests, P < 0.05 will be considered significant, and nonparametric testing will be applied where appropriate.

SECONDARY OUTCOMES:
Early Treatment Diabetic Retinopathy Study (ETDRS) Severity Level assessment of Clarus global, Optos global, and Standard 7 Field grading and statistical comparison | 1 day
  The images captured on each camera will be graded using the ETDRS severity scale. The total range of possible scores for severity level is from 10 (no DR) to 80 (PDR with vitreous hemorrhage); higher scores indicate increasing severity.
  Details of ETDRS severity scale: 10-No DR, 15-Probable DR, no MAs, 20-MAs only, 35-Mild NPDR, 43,47-Moderate NPDR, 53-Severe NPDR, 60-PDR status post scatter photocoagulation, 61,65,71-PDR, 80-PDR with vitreous hemorrhage, 90,95-Ungradable.
  ETDRS level agreement will be cross-tabulated and κ statistics calculated and assessed: <0.20, poor; 0.21-0.40, fair; 0.41-0.60, moderate; 0.61-0.80, substantial; and 0.81-1.00, almost perfect strength of agreement. Unweighted κ will be used to avoid potential bias by weighting. Agreement will also be tested for each severity level and k statistics analyzed.
Number of Ungradable ETDRS Images within the Clarus global, Optos global, and Standard 7 Field grading | 1 day
  The images captured within the global fields of the Clarus and Optos cameras and the 7 standard field image will be graded using the ETDRS severity scale. The proportion of ungradable images will be documented. On all tests, P < 0.05 will be considered significant, and nonparametric testing will be applied where appropriate.
Image quality assessment per image grader | 1 day
  The images captured on each camera for each participant will be assessed for quality using the Wisconsin Reading Center's 3-step confidence score. 1-High (image can be graded for both 7 field ETDRS and global severity level); 2-Adequate (image cannot be graded for global severity level); 3-Inadequate (image cannot be graded for ETDRS and global severity level).
Reason Image Quality is compromised per image grader | 1 day
  If Wisconsin Reading Center Confidence score of 2 or 3, a reason is selected (technical, patient, both patient and technical, unknown, or N/A). Eyes with photographs classified as ungradable will be excluded from agreement tables.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Blodi, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Health - University Station Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No